CLINICAL TRIAL: NCT07303699
Title: Population Pharmacokinetics and Pharmacodynamics of Standard First Line Anti-TB Versus Atorvastatin-Containing Regimens in the Treatment of Pulmonary Tuberculosis: A Sub-study of the ATORTUB Phase 2C Randomized Controlled Trial (ATORTUB popPK-PD Study)
Brief Title: ATORvastatin in Pulmonary TUBerculosis: a POPulation PharmacoKinetics -PharmacoDynamics Sub-study (ATORTUB popPK-PD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Obafemi Awolowo University Teaching Hospital (Other)
Collaborators: Open Philanthropy (Other); Obafemi Awolowo University (Other)
Responsible Party: Principal Investigator, Adewole Olufemi, Professor, Obafemi Awolowo University Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERC/2023/11/15/B; IRB/IEC/0004553 (Other: International)
Record Dates: First submitted 2025-09-21; First posted 2025-12-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Tuberculosis (TB)
Keywords: Pulmonary TB; Pulmonary Tuberculosis; Tuberculosis; Koch's disease; Mycobacterium tuberculosis; Isoniazid; Atorvastatin; Rifampicin; Rifampin; Ethambutol; pyrazinamide; Intensive Phase; Continuation Phase; statins; Antitubercular therapy (ATT)
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — Atorvastatin; Isoniazid; Protons; Pyrazinamide; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 20mg atorvastatin with standard of care (SOC) for TB (Experimental): Trial of 20mg atorvastatin with standard of care (SOC) for TB [2RHZE/4RH + 4AT(20)]
  Interventions: Drug: Atorvastatin 20 mg; Drug: Fixed dose combination of Rifampicin (R) Isoniazid (H) Pyrazinamid (Z) Ethambutol (E)
- 40mg atorvastatin with standard of care (SOC) for TB (Experimental): Trial of 40mg atorvastatin with standard of care (SOC) for TB [2RHZE/4RH + 4AT(40)]
  Interventions: Drug: Atorvastatin 40 mg; Drug: Fixed dose combination of Rifampicin (R) Isoniazid (H) Pyrazinamid (Z) Ethambutol (E)
- 60mg atorvastatin with standard of care (SOC) for TB (Experimental): Trial of 60mg atorvastatin with standard of care (SOC) for TB [2RHZE/4RH + 4AT(60)]
  Interventions: Drug: Atorvastatin 60 mg; Drug: Fixed dose combination of Rifampicin (R) Isoniazid (H) Pyrazinamid (Z) Ethambutol (E)
- standard of care (SOC) for TB (Active Comparator): Standard of Care (SOC) for TB [2RHZE/4RH]
  Interventions: Drug: Fixed dose combination of Rifampicin (R) Isoniazid (H) Pyrazinamid (Z) Ethambutol (E)

INTERVENTIONS:
Drug: Atorvastatin 20 mg — Participants will receive 16weeks of daily oral treatment with 20mg atorvastatin 4AT(20)]
  Other Names: Astin
  Arms: 20mg atorvastatin with standard of care (SOC) for TB
Drug: Atorvastatin 40 mg — Participants will receive 16 weeks of daily oral treatment with 40mg atorvastatin 4AT(40)]
  Other Names: Astin
  Arms: 40mg atorvastatin with standard of care (SOC) for TB
Drug: Atorvastatin 60 mg — Participants will receive 16weeks of daily oral treatment with 60mg atorvastatin 4AT(60)
  Other Names: Astin
  Arms: 60mg atorvastatin with standard of care (SOC) for TB
Drug: Fixed dose combination of Rifampicin (R) Isoniazid (H) Pyrazinamid (Z) Ethambutol (E) — Participants will receive 8 weeks of daily oral treatment with rifampin, isoniazid, pyrazinamide, ethambutol, followed by 16 weeks of daily treatment with rifampin, isoniazid [2RHZE/4RH]
  Other Names: Stop TB Kit

SUMMARY:
The purpose of this study is to assess pharmacokinetic parameters of atorvastatin at different doses when combined with the standard first line tuberculosis (TB) treatment regimen in adults with drug sensitive pulmonary TB. The pharmacokinetics parameters will be correlated with Pharmcodynamic measures and a PK/PD model that will identify an optimal dosing regimen of atorvastatin that is appropriate for the treatment of pulmonary tuberculosis will be developed.

DETAILED DESCRIPTION:
This is a pharmacokinetics-pharmacodynamics sub-study of ATORTUB trial (NCT06199921) and a dose finding study of atorvastatin in adults with pulmonary TB.

It is a parallel dose comparison trial in which participants will be randomised into four treatment arms. Participants in the experimental arms of the study will receive standard anti-TB therapy for 24 weeks plus oral atorvastatin daily in the first 16 weeks. Study participants will be followed up for another 6 months post treatment. Total study duration for participants will be 52 weeks post randomization, during which participants will attend several study visits. Sputum specimen collection, chest Xray, lung function test, and sparse pharmacokinetic sampling will be done at each visit.

The pharmacokinetic/ Pharmacodynamic data for atorvastatin will be used to identify a dose to be studied as adjunctive TB treatment in subsequent trials.

ELIGIBILITY:
Inclusion Criteria:

* Sputum specimen positive for tubercle bacilli on Gene Xpert or direct smear microscopy
* Either no previous anti-TB chemotherapy, or less than 2 weeks of previous chemotherapy
* Aged 12years and above
* A firm home address that is readily accessible for visiting
* Agreement to participate in the study and to give a sample of blood for HIV testing
* Normal baseline laboratory values at or within 14 days prior to screening:

  * Serum or plasma alanine aminotransferase (ALT) less than or equal to 3 times the upper limit of normal
  * Serum or plasma total bilirubin less than or equal to 2.5 times the upper limit of normal
  * Serum or plasma creatinine level less than or equal to 2 times the upper limit of normal
  * Serum or plasma potassium level greater than or equal to 3.5 meq/L
  * Hemoglobin level of 7.0 g/dL or greater
  * Platelet count of 100,000/mm3 or greater
* Informed consent to participate in the study and to give a sample of blood for HIV testing

Exclusion Criteria:

* Participants known or suspected of having any form of drug resistance TB.
* Patients co infected with HIV
* Those with poor general condition where no delay in treatment can be tolerated
* Evidence of clinically significant metabolic or co morbid medical conditions ; malignancy; or other diseases like history of or current cardiovascular disorder such as heart failure, coronary heart disease, arrhythmia.
* Known or family history of bleeding disorders.
* Any renal impairment characterized by serum creatinine clearance of 1.5 x upper limit of normal of the clinical laboratory reference range at screening.
* Myositis and or Creatinine phosphokinase three times upper limit of normal
* Patient in a moribund state
* Has TB meningitis
* Presence of any of the pre-existing non-TB diseases outlined in the protocol
* Diabetes mellitus
* Hypertension
* Currently on anti TB medication
* Any other chronic illness/ co morbidities that warrants being on daily routine medications
* Presence of a psychiatric illness
* pregnant, or breast feeding mothers
* Current Tobacco Smokers/ tobacco use in any form
* Alcoholism
* alcoholic beverages, food or drinks containing methyl- xanthine (i.e. energy drinks, tea leaves, coffee beans, cocoa, kola nuts, medications e.g. theophylline). Ingestion of grapefruit/ products containing grapefruit juice, bitter oranges, garlic supplements, St John's Wort or other herbal supplements, within 7 days prior to the first treatment and throughout the study will not be allowed.
* Individuals that are enrolled in other therapeutic clinical trials

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-03 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC 0-24) for atorvastatin acid, rifampicin, isoniazid and their metabolites at steady state | Sampling will be on day 14 & week 8, 16 and 24 post randomization
  Sparse pharmacokinetic sampling will be employed during participants treatment follow up visits for the determination of plasma concentrations of atorvastatin acid, rifampicin, isoniazid. and their active metabolites (2-hydroxyl atorvastatin 4- hydroxyl atorvastatin, acetyl - isoniazid, desacetyl - rifampicin). AUC will be estimated using Population Pharmacokinetics analysis
Peak Plasma Concentration (Cmax) for atorvastatin acid, rifampicin, isoniazid and their metabolites at steady state | Sampling will be on day 14 & week 8, 16 and 24 post randomization
  Sparse pharmacokinetic sampling will be employed during participants treatment follow up visits for the determination of plasma concentrations of atorvastatin acid, rifampicin, isoniazid. and their active metabolites (2-hydroxyl atorvastatin 4- hydroxyl atorvastatin, acetyl - isoniazid, desacetyl - rifampicin). Cmax will be estimated using Population Pharmacokinetics analysis
Plasma Clearance (Cl/F) in mL/min of atorvastatin acid, rifampicin, isoniazid and their metabolites at steady state | Sampling will be on day 14 & week 8, 16 and 24 post randomization
  Sparse pharmacokinetic sampling will be employed during participants treatment follow up visits for the determination of plasma concentrations of atorvastatin acid, rifampicin, isoniazid. and their active metabolites (2-hydroxyl atorvastatin 4- hydroxyl atorvastatin, acetyl - isoniazid, desacetyl - rifampicin). Plasma clearance of aforementioned drugs and metabolites will be estimated using Population Pharmacokinetics analysis

SECONDARY OUTCOMES:
Correlation between AUC 0-24 of atorvastatin acid, 2-hydroxyl atorvastatin and 4- hydroxyl atorvastatin at steady state and days 0-14 early bactericidal activity in participants on atorvastatin-based regimens | day 14 post randomization
  steady state AUC 0-24 of atorvastatin acid, 2-hydroxyl atorvastatin and 4- hydroxyl atorvastatin will be correlated with early bactericidal activity on day 14. Early bactericidal activity will be measured as the daily rate of change in log10 Colony Forming Units of M. Tuberculosis in Sputum on Solid Media
Correlation between Cmax of atorvastatin acid, 2-hydroxyl atorvastatin and 4- hydroxyl atorvastatin at steady state and days 0-14 early bactericidal activity in participants on atorvastatin-based regimens | day 14 post randomization
  Cmax of atorvastatin acid, 2-hydroxyl atorvastatin and 4- hydroxyl atorvastatin will be correlated with early bactericidal activity on day 14. Early bactericidal activity will be measured as the daily rate of change in log10 Colony Forming Units of M. Tuberculosis in Sputum on Solid Media
Correlation between Cmax of atorvastatin acid, 2-hydroxyl atorvastatin and 4- hydroxyl atorvastatin at steady state and time to stable sputum culture conversion | 2 - 24 weeks post randomization
  Time to achieve culture negative sputum result as measured by growth on solid mycobacteria culture medium
Correlation between AUC 0-24 of atorvastatin, atorvastatin acid, 2-hydroxyl atorvastatin and 4- hydroxyl atorvastatin) at steady state and change in baseline chest Xray severity score at 4, 6 and 12 months | 16 -52weeks post randomisation
  Change in baseline chest Xray severity score as measured by Timika Chest X ray scoring system. At least 30% reduction in Chest x-ray severity score is desirable
Correlation between AUC 0-24 of atorvastatin acid, 2-hydroxyl atorvastatin and 4- hydroxyl atorvastatin at steady state and time to stable sputum culture conversion | 2 - 24 weeks post randomization
  Time to achieve culture negative sputum result as measured by growth on solid mycobacteria culture medium
Correlation between Cmax of atorvastatin, atorvastatin acid, 2-hydroxyl atorvastatin and 4- hydroxyl atorvastatin) at steady state and change in baseline chest Xray severity score at 4, 6 and 12 months | 16 - 52 weeks post randomization
  Change in baseline chest Xray severity score as measured by Timika Chest X ray scoring system. At least 30% reduction in Chest x-ray severity score is desirable
Correlation between AUC 0-24 of atorvastatin acid, 2-hydroxyl atorvastatin and 4- hydroxyl atorvastatin) at steady state and change in baseline lung function at 4, 6 and 12 months | 16 -52 weeks post randomization
  Change in baseline lung function (FEV1 and FVC) test will be assessed using a spirometer at 4, 6 and 12 months. At least 15% improvement in FEV1 and FVC is desirable.
Correlation between Cmax of atorvastatin acid, 2-hydroxyl atorvastatin and 4- hydroxyl atorvastatin) at steady state and change in baseline lung function at 4, 6 and 12 months | 16 - 52 weeks post randomization
  Change in baseline lung function (FEV1 and FVC) test will be assessed using a spirometer at 4, 6 and 12 months. At least 15% improvement in FEV1 and FVC is desirable.
The optimal dose of atorvastatin that will be safe and effective as an adjunctive pulmonary TB treatment | week 52 post randomization
  A pharmackinetic - Pharmacodynamic (PK/ PD) model will be developed for each drug (using PK -PD data generated from other secodary outcomes described above) and the the optimal dose of atorvastatin that will be appropriate as adjunctive TB treatment will be investigated using Monte-Carlo simulations.

CONTACTS AND LOCATIONS:
Overall Officials: Olanisun O Adewole, MD, Principal Investigator — Obafemi Awolowo University / Teaching Hospital, Ile Ife, Nigeria; Bolanle A Omotoso, MD, Study Director — Obafemi Awolowo University /Teaching Hospital, Ile- Ife, Osun State, Nigeria; Olanisun O Adewole, MD, Study Chair — Obafemi Awolowo University /Teaching Hospital, Ile- Ife, Osun State, Nigeria
Locations (3):
- Nigeria (3):
  - National Tuberculosis and Leprosy Training Centre, Saye, Zaria, Kaduna State
  - Federal Teaching Hospital, Katsina, Katsina State
  - Obafemi Awolowo University Teaching Hospitals Complex, Ile Ife, Osun state, Nigeria, Ile-Ife, Osun State

IPD SHARING:
Plan to Share IPD: No